CLINICAL TRIAL: NCT01130623
Title: A Phase I Study of Pazopanib as a Single Agent for Children With Relapsed or Refractory Solid Tumors, Including CNS Tumors
Brief Title: A Phase I Study of Pazopanib as a Single Agent for Children With Refractory Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: CTEP/National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100120; 10-C-0120
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-11-18

CONDITIONS: Sarcoma; Neuroblastoma; Wilms Tumor; Osteosarcoma; Brain Tumor
Keywords: VEGF Inhibitor; Maximum Tolerated Dose; Dose Escalation; Pharmacokinetics; Antitumor Activity; Pediatric Cancer; Solid Tumor; Sarcoma; Neuroblastoma; Wilms Tumor; Osteosarcoma; Brain Tumor
MeSH Terms: conditions — Sarcoma; Neuroblastoma; Wilms Tumor; Osteosarcoma; Brain Neoplasms; Neoplasms | interventions — pazopanib

INTERVENTIONS:
Drug: Pazopanib (GW786034)

SUMMARY:
Background:

- Pazopanib, a drug that inhibits the growth of new blood vessels in tumors, was recently approved by the Food and Drug Administration to treat advanced kidney cancer in adults. Pazopanib has been used in only a small number of adults, and more research is needed on whether it is safe and effective to use in children. Researchers are interested in determining safe and effective treatment doses of pazopanib in children, and in other studies will examine which form of pazopanib treatment (tablet or liquid) is most effective and well tolerated.

Objectives:

* To determine a safe and effective dose of pazopanib to treat solid tumors in children.
* To study the effects of pazopanib on blood cells, blood flow, and human development.

Eligibility:

- Children, adolescents, and young adults between 1 and 21 years of age who have been diagnosed with solid tumors that have not responded to treatment.

Design:

* Eligible participants will be screened with a physical examination, blood and tumor samples, and imaging studies.
* Participants will receive pazopanib tablets for 28-day cycles of treatment. Pazopanib should be taken on an empty stomach, at least 1hour before or 2 hours after a meal. Participants may receive pazopanib for up to 24 cycles unless the tumor does not respond or participants develop serious side effects.
* Blood samples will be taken on days 1, 15, 22, and 27 of the first cycle of pazopanib, with additional samples taken every 8 weeks during subsequent cycles.
* An optional part of the study will collect additional blood samples at regular intervals for 24 hours after the first dose of pazopanib and at regular intervals after another dose during the second or third week of the first treatment cycle.

DETAILED DESCRIPTION:
Background:

* Pazopanib is a potent and selective multi-target receptor tyrosine kinase inhibitor of vascular endothelial growth factor (VEGF) receptors (VEGFR)-1, -2, and -3, c-kit and platelet derived growth factor (PDGF) receptors-alpha and -beta.
* Preclinical experiments demonstrate that pazopanib causes significant and dose-dependent inhibitory effects on cell proliferation and inhibition of VEGF-induced VEGFR-2 phosphorylation, growth inhibition of a variety of human tumor xenografts in mice, and inhibition of basic fibroblast growth factor-(bFGF) and VEGF-induced angiogenesis in murine models.
* Pazopanib has been evaluated in adult subjects with solid tumors in Phase I and II studies, and objective anti-tumor activity has been observed in a variety of tumor types.

Objectives:

Primary Objectives:

* To estimate maximum tolerated dose (MTD) and/or recommended Phase II dose of oral pazopanib administered on a once daily schedule to children with refractory solid tumors.
* To define the toxicities of oral pazopanib administered as either a tablet or suspension.
* To characterize the pharmacokinetics of oral pazopanib in children with refractory solid tumors.

Secondary Objectives:

* To preliminarily define the antitumor and biologic activity of oral pazopanib, and to explore the changes in tumor vascular permeability following initiation of pazopanib.
* To preliminarily assess VEGF haplotype/phenotype relationships in children with cancer.
* To explore pazopanib concentration-effect relationships with biomarkers and with clinical outcomes.

Eligibility:

* Part 1 (Phase I Dose Escalation) and 2a (Suspension Formulation Component):

  --Patients greater than 12 months and less than or equal to 21 years of age with measureable or evaluable relapsed or refractory solid tumors including CNS tumors with histologic verification except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevation of tumor markers.
* Part 2b (Expanded Imaging Cohort):

  --Patients greater than 2 years and less than or equal to 25 years of age with histologically verified relapsed or refractory soft tissue sarcoma, desmoplastic small round cell tumor or extraosseus Ewing sarcoma with measurable disease (greater than or equal to 2 cm) in the head, neck, extremity or fixed within the thorax, abdomen or pelvis.
* Performance score: Karnofsky greater than or equal to 50% for patients 16 years of age; Lansky greater than or equal to 50 for patients less than or equal to 16 years of age.
* Must have fully recovered from acute toxic effects from all prior therapy which have been completed within the specified prior time frame. Have adequate organ function as determined by laboratory evaluation.

Design:

* This is a rolling six phase I trial design of pazopanib administered orally once daily continuously on a 28 day cycle.
* Therapy may continue for up to 24 cycles in the absence of progressive disease or unacceptable toxicity.
* Part 1 is the phase I dose escalation portion (Completed). Once the MTD or phase II recommended dose is defined, up to 16 additional patients will enroll in Part 2a to obtain safety and pharmacokinetic data for the suspension formulation. In addition, up to 10 patients with recurrent/refractory soft tissue sarcoma and a measurable lesion will be enrolled in Part 2b at the MTD or recommended Phase II dose to further explore changes in tumor vascular permeability using dynamic contrast enhanced MRI.
* Participation in correlative biology studies or pharmacokinetic studies will be optional in Part 1; pharmacokinetic studies will be required in Part 2a; and imaging and limited pharmacokinetic sampling will be required in Part 2b.

ELIGIBILITY:
* Eligibility:
* Part 1 (Phase I Dose Escalation) and 2a (Suspension Formulation Component):

  --Patients greater than 12 months and less than or equal to 21 years of age with measureable or evaluable relapsed or refractory solid tumors including CNS tumors with histologic verification except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevation of tumor markers.
* Part 2b (Expanded Imaging Cohort):

  --Patients greater than 2 years and less than or equal to 25 years of age with histologically verified relapsed or refractory soft tissue sarcoma, desmoplastic small round cell tumor or extraosseus Ewing sarcoma with measurable disease (greater than or equal to 2 cm) in the head, neck, extremity or fixed within the thorax, abdomen or pelvis.
* Performance score: Karnofsky greater than or equal to 50% for patients 16 years of age; Lansky greater than or equal to 50 for patients less than or equal to 16 years of age.
* Must have fully recovered from acute toxic effects from all prior therapy which have been completed within the specified prior time frame. Have adequate organ function as determined by laboratory evaluation.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05-10; Primary Completion 2011-11-18 (Actual); Study Completion 2011-11-18 (Actual)

PRIMARY OUTCOMES:
To estimate MTD and Phase II dose of oral pazopanib.
To define the toxicities of oral pazopanib tablet or suspension.
To characterize PKs.

SECONDARY OUTCOMES:
To define antitumor and biologic activity and explore changes in tumor vascular permeability. To assess VEGF haplotype/phenotype relationships and explore concentration-effect with biomarkers and clinical outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hanahan D, Weinberg RA. The hallmarks of cancer. Cell. 2000 Jan 7;100(1):57-70. doi: 10.1016/s0092-8674(00)81683-9. No abstract available. PMID 10647931
- [Background] Bigler SA, Deering RE, Brawer MK. Comparison of microscopic vascularity in benign and malignant prostate tissue. Hum Pathol. 1993 Feb;24(2):220-6. doi: 10.1016/0046-8177(93)90304-y. PMID 8432518
- [Background] Bochner BH, Cote RJ, Weidner N, Groshen S, Chen SC, Skinner DG, Nichols PW. Angiogenesis in bladder cancer: relationship between microvessel density and tumor prognosis. J Natl Cancer Inst. 1995 Nov 1;87(21):1603-12. doi: 10.1093/jnci/87.21.1603. PMID 7563203